CLINICAL TRIAL: NCT01870050
Title: A Double-blind, Randomized, Parallel-group, Side-by-side Single-center Study Comparing a Topical Steroid / Vehicle Combination to a Topical Steroid / Topical Dapsone Combination in Patients With Lichen Simplex Chronicus and/or Prurigo Nodularis
Brief Title: Dapsone Prurigo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Joerg Albrecht, Attending Physician, Cook County Health
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cookderm 01
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Lichen Simples Chronicus and Prurigo
Keywords: lichen simplex chronicus; prurigo
MeSH Terms: conditions — Prurigo; Neurodermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dapsone gel - verum (Active Comparator): dapsone gel - verum
  Interventions: Drug: Dapsone gel - verum
- dapsone gel - vehicle only (Placebo Comparator)

INTERVENTIONS:
Drug: Dapsone gel - verum
  Other Names: aczone gel
  Arms: dapsone gel - verum

SUMMARY:
Principal aim of this study is to assess whether a combination of topical dapsone and clobetasol as a topical steroid is superior to clobetasol alone as treatment of prurigo nodularis or lichen simplex chronicus in a side to side comparison. The study is primarily exploratory and essentially meant to inform the sponsor whether further development of a combination treatment formulation is warranted

ELIGIBILITY:
Inclusion Criteria:

* • Active prurigo nodularis or lichen simplex chronicus - diagnosed by clinical exam

  * For lichen simplex chronicus patients: Severity of maximum pruritus in the last 24 hrs at least 5 out of 10 on a visual analogue scale.
  * For prurigo nodularis patients: Excoriations or signs of other scratch related activity at presentation to demonstrate active disease
  * Symmetrical disease/excoriations allowing for a side-by-side comparison (eg, bilateral lichen simplex chronicus or bilateral prurigo nodularis) - genitals, face, axillae or neck cannot be used for side-to-side comparison
  * Willing to refrain from use of all other topical medications in the treatment areas.
  * Able and willing to provide written informed consent
  * Willing and able to understand and comply with the requirements of the study, apply the treatment combinations as instructs, attend required study visits, comply with study prohibitions and able to complete the study.
  * Male or non-preganant, non-lactating female between 18 and 75 years of age, inclusive
  * For females of child-bearing potential, willing to use adequate birth control during the study conduct

Exclusion Criteria:

* • History of non-compliance with follow up visits

  * Should we exclude failure to certain treatments as an exclusion criterion? Patients who failed oral dapsone should be excluded
  * Presence of any skin condition on the treatment areas that would interfere with the diagnosis or assessment of active lichen simplex chronicus and/or prurigo nodularis (eg, rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis or bacterial folliculitis)
  * Excessive hair in the treatment area that would interfere with diagnosis or assessment of lichen simplex chronicus and/or prurigo nodularis
  * History of hypersensitivity or allergy to topical steroids, dapsone, or any other treatment product components
  * Use of tanning booths, sunbathing or excessive exposure to the sun during the study
  * Consumes excessive amount of alcohol, abuses drugs, or has any condition that would compromise compliance with this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Pruritus based on visual analogue scale in side to side comparison | 8 weeks

SECONDARY OUTCOMES:
5 D itch scale in side to side comparison | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Albrecht, MD, Principal Investigator — J.H.Stroger Hospital of Cook County
Locations (1):
- J H Stroger Hospital of Cook County, Chicago, Illinois, United States